CLINICAL TRIAL: NCT04618640
Title: A Multicenter, Single-group, Phase III Study to Evaluate the Immunogenicity and Safety of DTaP-IPV Vaccine Administered as a Boosting Dose to Healthy Children of 4-6 Years Who Completed the Primary Vaccination Against Diphtheria, Tetanus, Pertussis, and Poliomyelitis by Participating in the Phase III Study, BR-DTPP-CT-301, or by Receiving Routine Vaccination
Brief Title: To Evaluate the Immunogenicity and Safety of DTaP-IPV Vaccine Administered as a Boosting Dose to Healthy Children of 4-6 Years
Acronym: Aladdin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boryung Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BR-DTPP-CT-302
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis
Keywords: DTaP-IPV; Boosting Dose
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis

STUDY DESIGN:
Intervention Model Description: DTaP-IPV combined vaccine, 0.5mL, imtramuscular
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTaP-IPV combination vaccine (Experimental): DTaP-IPV 0.5ml IM boosting
  Interventions: Biological: DTaP-IPV combination vaccine

INTERVENTIONS:
Biological: DTaP-IPV combination vaccine — Dosage and administration: A single intramuscular injection of 0.5 mL will be given to healthy children aged 4 to 6 years

SUMMARY:
The study objective is to assess the immunogenicity and safety of DTaP-IPV combination vaccine administered as a boosting dose to healthy 4 to 6-year-old children who received three doses of primary immunization against diphtheria, tetanus, pertussis, and polio.

ELIGIBILITY:
Inclusion Criteria:

1. A subject's parent/legal representative provides a written consent after being informed about the study objective, methods, effect of the study vaccine, and other relevant information
2. Documented record of the three doses of primary immunization against diphtheria, tetanus, pertussis, and polio either by participating in the previous study, BR-DTPP-CT-301 or by following the national immunization schedule under usual clinical setting (the primary immunization should have been initiated after 6 weeks of age and at minimal interval of 4 weeks)
3. Receipt of a boosting dose against diphtheria, tetanus, and pertussis until 2 years of age; therefore, total of four vaccination records against diphtheria, tetanus, and pertussis and three against polio
4. Healthy male or female children, aged 4 to 6 years on the day of the vaccination

Exclusion Criteria:

1. Children aged 7 years or older
2. Previously received DTaP vaccine five times or more, including the doses received in the BR-DTPP-CT-301 study, either by a combination vaccine or a separate vaccine
3. Previously received IPV vaccine four times or more, including the doses received in the BR-DTPP-CT-301 study, either by a combination vaccine or a separate vaccine
4. The fourth dose of DTaP vaccine was postponed and administered after 4 years of age
5. Acute febrile illness with fever ≥ 38.0°C (tympanic) on the day of the vaccination
6. Moderate to severe systemic acute illness with or without fever
7. History of diphtheria, tetanus, pertussis, or polio (poliomyelitis)
8. Dysfunctional immune system or congenital or acquired immunodeficiency
9. Had encephalopathy of unknown etiology within 7 days following a previous dose of DTaP vaccine
10. Received a vaccine other than the protocol-permitted vaccines within 28 days from the study vaccination day or are planned to receive such a vaccine during the study period
11. Received systemic corticosteroid treatment at immunosuppressive dosage within 28 days from the study vaccination day or are planned to receive such a treatment during the study period (exceptionally, administration of prednisolone ≤ 0.5 mg/kg/day for up to 14 continuous days is allowed)
12. Received immunoglobulins or blood products within 90 days before the study vaccination day or are planned to receive such products during the study period
13. Had severe allergic reaction (e.g. anaphylaxis) to ingredients of the investigational product or bears such a possibility
14. Currently enrolled in another clinical trial or planned to participate in another clinical trial
15. Any other reasons that preclude the eligibility of the subject, based on investigator's decision

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate after boosting vaccination | boosting vaccination after Day 28 [+14 days]
  Antibodies will be measured by enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Seroprotection rate for anti-DT, anti-TT, and anti-poliovirus or seropositive (>30 IU/mL) rate for anti-PT and anti-FHA before boosting vaccination | Day 1 Pre-vaccination
  Seroprotection rate
Minimal seroprotection rate for anti-DT and anti-TT (≥ 0.01 IU/mL) before boosting vaccination | Day 1 Pre-vaccination
  Seroprotection rate (≥ 0.01 IU/mL)
Pre-booster antibody level | Day 1 Pre-vaccination
Post-booster antibody level | boosting vaccination after Day 28 [+14 days]
Geometric mean ratio (GMR) between the pre- and post-booster antibody level | Day 1 Pre-vaccination and boosting vaccination after Day 28 [+14 days]
GMR between the pre- and post-booster antibody level in each subgroup depending on the pre-booster antibody level (≥ seroprotective/seropositive level or < seroprotective/seropositive level) | Day 1 Pre-vaccination and boosting vaccination after Day 28 [+14 days]
Reverse cumulative distribution curves for pre- and post-booster antibody level | Day 1 Pre-vaccination and boosting vaccination after Day 28 [+14 days]
Seroprotection rate for anti-DT, anti-TT, and anti-poliovirus or seropositive (>30 IU/mL) rate for anti-PT and anti-FHA after boosting vaccination | boosting vaccination after Day 28 [+14 days]
Proportion of subjects with post-booster antibody levels for anti-DT and anti-TT ≥1.0 IU/mL | boosting vaccination after Day 28 [+14 days]

CONTACTS AND LOCATIONS:
Overall Officials: Byeonguk Eun, Study Chair — Eulji University Hospital
Locations (26):
- South Korea (26):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Medical Center, Anyang
  - Changwon Fatima Hospital, Changwon
  - KeiMyung University Dongsan Medical Center, Daegu
  - Hallym University Medical Center, Gyeonggi-do
  - Myongji Hospital, Gyeonggi-do
  - Wonkwang University Hospital, Iksan
  - Inha University Hospital, Incheon
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Mediplex Sejong Hospital, Sejong
  - Bundang Cha Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Eulji University Hospital, Seoul
  - Gangnam Sevrance Christian Hospital, Seoul
  - Hanil General Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - KyungHee University Hospital at Gangdong, Seoul
  - KyungHee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - Wonju Sevrance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No